CLINICAL TRIAL: NCT02698748
Title: Evaluating the Potential Role of Chloroquine in Preventing Infections During Elimination Campaigns: A Randomized, Single-blind, Placebo-controlled Trial in Asymptomatic Mozambican Adults
Brief Title: Evaluating the Role of Chloroquine for Malaria Elimination
Acronym: Cloroquina
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centro de Investigacao em Saude de Manhica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CNBS (173/CNBS/13)
Record Dates: First submitted 2015-01-13; First posted 2016-03-04 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2016-02

CONDITIONS: Malaria
Keywords: Chloroquine; Malaria Elimination; P.falciparum; Clinical Trial; Mozambique; Adults
MeSH Terms: conditions — Malaria | interventions — Chloroquine; chloroquine diphosphate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chloroquine (Experimental): Chloroquine sulphate (Meriquine®; 250mg; 150 mg of chloroquine base; Baroda, India) will be administered at a total dose of 25 mg/kg (expressed as mg of CQ base per kg body weight, once daily during 3 consecutive days, following the schedule 10mg/kg Day 1; 10mg/kg day 2 and 5 mg/kg day 3).
  Interventions: Drug: Chloroquine
- Placebo (Placebo Comparator): Placebo pills will be standard placebo capsules filled with powder contents with no pharmaceutical activity. They will not be identical to the chloroquine tablets, so the study will not be double blind, but rather single blinded. Placebo tablets will be manufactured by the pharmaceutical department of the Hospital Clínic, in Barcelona, Spain.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chloroquine — Chloroquine sulphate (Meriquine®; 250mg; 150 mg of chloroquine base; Baroda, India) will be administered at a total dose of 25 mg/kg (expressed as mg of CQ base per kg body weight, once daily during 3 consecutive days, following the schedule 10mg/kg Day 1; 10mg/kg day 2 and 5 mg/kg day 3).
  Other Names: Chloroquine Phosphate
  Arms: Chloroquine
Drug: Placebo — Placebo Placebo pills will be standard placebo capsules filled with powder contents with no pharmaceutical activity. They will not be identical to the chloroquine tablets, so the study will not be double blind, but rather single blinded. Placebo tablets will be manufactured by the pharmaceutical department of the Hospital Clínic, in Barcelona, Spain
  Other Names: Placebo capsules
  Arms: Placebo

SUMMARY:
One of the proposed ideas for malaria elimination includes the use of drugs to interrupt malaria transmission by exhausting the human reservoir of infection. Theoretically, mass treatment of an entire population with a very effective and rapid-acting drug (for instance an ACT), followed by the administration of an effective prophylactic regime during a minimum of four weeks, so as to outlast the typical development period of Plasmodium parasites in Anopheline mosquitoes, could achieve the same objective. In this respect, chloroquine (CQ) would be an appropriate candidate. This drug exhibits two conditions that make it attractive for elimination campaigns: 1) It has been demonstrated to have an excellent safety profile, allowing for its use in all age groups including pregnant women and children; and 2) Its relatively long elimination half life (t1/2=1-2 months) can provide a long post-treatment prophylactic effect. Recent evidence suggests that CQ sensitivity may be returning in places where discontinuation has reduced the drug pressure to the parasite populations. In countries such as Malawi, P. falciparum seems to have regained full sensitivity to CQ, and molecular markers of antiCQ resistance have nearly disappeared. While this does not support the reintroduction of CQ as first line therapy, it does suggest that, if proven sensitive in a given area, it could play a prophylactic role in malaria elimination strategies when used in combination with other drugs or tools. Thus, we intend to evaluate the potential role of chloroquine in preventing infections during elimination campaigns by performing a randomized, single-blind, placebo-controlled trial in asymptomatic Mozambican adults.

Choosing asymptomatic parasitaemic adult males from a malaria-endemic area as our study population introduces limited risks when administering a drug with an uncertain efficacy (47% efficacious in 2001-2002). In malaria-endemic areas, this age group has a remarkably low risk of developing severe disease (irrespective of clinical symptoms), and it is foreseeable that parasitemia may be well tolerated, and in certain cases, spontaneously cleared from the individual's blood as a result of the immune system. In the unlikely event of any clinical symptomatology appearing throughout the follow-up, individuals will be examined by a study clinician and treated immediately with the country's first-line malaria treatment (artemether-lumefantrine, Coartem ®).

DETAILED DESCRIPTION:
This surveillance study is a two-arm prospective evaluation of parasitological responses to directly observed treatment with CQ (vs. placebo) for the clearing of asymptomatic parasitemia. People with asymptomatic P. falciparum parasitaemia, defined as the presence of a P. falciparum infection in the absence of any clinical symptomatology including fever, history of fever in the preceding 24 hours, malaise, fatigue, chills, or any other symptoms that may be derived from the malarial infection, who meet the study inclusion criteria will be enrolled, treated on site with CQ phosphate (25mg/Kg CQ base divided in three daily doses: 10mg/kg day 1 (usually 4 tablets); 10mg/kg day 2 (4 tablets) and 5mg/kg day 3 (2 tablets)) or placebo pills (same schedule, 4 tablets day one and two; and 2 tablets on day three), and monitored for 28 days. The follow-up will consist of a fixed schedule of check-up visits and corresponding clinical and laboratory examinations. On the basis of the results of these assessments, the patients will be classified as having therapeutic failure (early or late) or an adequate response. The proportion of patients experiencing therapeutic failure during the follow-up period will be used to estimate the efficacy of the study drug. PCR analysis will be used to distinguish between a true recrudescence due to treatment failure and episodes of reinfection.

ELIGIBILITY:
Inclusion Criteria:

* Male individuals
* P. falciparum infection detected by microscopy (Minimum 250 parasites/microliter; Maximum 10.000parasites/microliter)
* Ability to swallow oral medication
* Ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule; and
* Informed consent from the participant individual

Exclusion Criteria:

* Age <18 years
* Female individuals
* Axillary temperature >=37.5ºC
* Presence of any other co-existing clinical condition that in the opinion of the recruiting physician would not allow the individual to be considered a "healthy" asymptomatic carrier
* Regular medication which may interfere with antimalarial efficacy or antimalarial pharmacokinetics, such as Cotrimoxazole
* History of hypersensitivity reactions or contraindications to CQ
* Known HIV positive patients in treatment with antiretrovirals

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Adequate parasitologic response (APR) to therapy | 28 days after first day of drug intake
  the absence of parasitemia at the end of the trial's follow-up period (Day 28), regardless of axillary temperature, without having previously met any of the criteria for early and late treatment failure

SECONDARY OUTCOMES:
Early parasitologic failure | 1-3 days after first day of drug intake
  Detection of parasites once the initial parasitemia has been cleared in the time period from day 1 to day 3 after first day of drug intake
Late parasitologic failure | 4-28 days after first day of drug intake
  The detection of parasites in patients having cleared their initial parasitemia anytime from day 4 to day 28
Prevalence of chloroquine conferring pfcrt K76T mutation in pre-treatment infections | 0 days after first day of drug intake
  Proportion of the isolates detected with this specific mutation among isolates at baseline (before study drug initiation)
Rates of pre treatment pfcrt K76T mutation in cases of chloroquine treatment failure | 0 days after first day of drug intake
  Proportion of the isolates detected with this specific mutation at baseline among cases with confirmed treatment failure those
Rates of post treatment pfcrt K76T mutation in cases of chloroquine treatment failure | 28 days after first day of drug intake
  Proportion of the isolates detected as new infections or recrudescent ones with this specific mutation
Clearance time of parasitaemia | 28 days after first day of drug intake
  time in hours until the clearance of parasitemia

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Aide, MD, MSc, PhD, Principal Investigator — Centro de Investigação em Saude de Manhiça
Locations (1):
- Centro de Investigaçao em Saude de Manhiça, Manhiça, Maputo Province, Mozambique

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Galatas B, Marti-Soler H, Nhamussua L, Cistero P, Aide P, Saute F, Menendez C, Rabinovich NR, Alonso PL, Bassat Q, Mayor A. Dynamics of Afebrile Plasmodium falciparum Infections in Mozambican Men. Clin Infect Dis. 2018 Sep 14;67(7):1045-1052. doi: 10.1093/cid/ciy219. PMID 29546346
- [Derived] Galatas B, Nhamussua L, Candrinho B, Mabote L, Cistero P, Gupta H, Rabinovich R, Menendez C, Macete E, Saute F, Mayor A, Alonso P, Bassat Q, Aide P. In-Vivo Efficacy of Chloroquine to Clear Asymptomatic Infections in Mozambican Adults: A Randomized, Placebo-controlled Trial with Implications for Elimination Strategies. Sci Rep. 2017 May 2;7(1):1356. doi: 10.1038/s41598-017-01365-4. PMID 28465550